CLINICAL TRIAL: NCT04880161
Title: A Randomized, Double-Blinded, Placebo-Controlled Phase I Study to Evaluate the Safety and Efficacy of Ampion in Patients With Prolonged Respiratory Symptoms Due to COVID-19 (Long COVID)
Brief Title: A Study to Evaluate Ampion in Patients With Prolonged Respiratory Symptoms Due to COVID-19 (Long COVID)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-018
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — aspartyl-alanyl-diketopiperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Ampion
  Interventions: Biological: Ampion
- Control (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ampion — Inhaled Ampion
  Arms: Active
Other: Placebo — Inhaled Placebo
  Arms: Control

SUMMARY:
This is a phase I study to evaluate the safety and efficacy of inhaled Ampion on patients with prolonged respiratory symptoms due to COVID-19 (Long COVID).

DETAILED DESCRIPTION:
Increasing numbers of people with COVID-19 are experiencing the lingering effects of COVID-19 and continue to have prolonged respiratory complications months after the onset of the disease, also known as Post-Acute Sequelae of SARS-CoV-2 (PASC), long-COVID, and/or long-hauler patients.

The SARS-CoV-2 virus is transmitted through the respiratory system, which can cause a severe dysregulation of the immune response and damage in the lungs. Chronic, prolonged inflammation of the lungs maybe responsible for a myriad of continuing respiratory signs and symptoms post-infection, including cough, shortness of breath, chest discomfort, low exercise tolerance and low blood oxygen saturation.

Ampion is the low molecular weight filtrate of human serum albumin with the in vitro ability to modulate inflammatory cytokine levels. Ampion has the potential to improve clinical outcomes for long-COVID patients.

This study aims to evaluate the safety of Ampion and the clinical outcomes in patients with long-COVID.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults: ≥ 18 years.
2. Must have a clinical diagnosis of COVID-19 at least 4 weeks prior to the screening date, with at least one of clinical symptoms (e.g., fever ≥ 38°C, fatigue, cough) and a positive result by the reverse-transcription polymerase chain reaction (RT-PCR) testing or equivalent.
3. Experiencing at least two COVID-19 respiratory symptoms with a score of two or higher using the FDA Assessment of 14 Common COVID-19-Related Symptoms questionnaire for at least 4 weeks (28 days) after initial positive COVID-19 diagnosis: cough, sore throat, runny/stuffy nose, shortness of breath (difficulties breathing), tightness of chest, low exercise tolerance.
4. Able to bear weight and ambulate a minimum of 10 meters distance.
5. Women of childbearing potential and their partner must agree to use at least one highly effective method of contraception (e.g., hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], intrauterine devices, bilateral tubal occlusion, or sexual abstinence) for the duration of the study.
6. Informed consent obtained from the patient or the patient's legal representative.

Exclusion Criteria:

1. Subjects who require hospitalization.
2. Patient has severe chronic obstructive or restrictive pulmonary disease (COPD) as defined by prior pulmonary function tests, chronic renal failure, or significant liver abnormality (e.g., cirrhosis, transplant, etc.).
3. History of Chronic Fatigue Syndrome prior to COVID-19 infection.
4. Patient is on chronic immunosuppressive medication.
5. Patient requires surgery that could be life-threatening within the study window.
6. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion) or ingredients in 5% human albumin (N-acetyl tryptophan, sodium caprylate).
7. Patient has known pregnancy or is currently breastfeeding.
8. Participation in a trial such that enrollment in this study would fall within the time frame of the half-life of the other investigational product(s).
9. Clinically significant findings via electrocardiogram (ECG), including acute myocardial infarction, acute ischemic changes, atrial fibrillation, atrial flutter, paced rhythms in individuals who have undergone permanent pacemaker placement, evidence of prior infarction, unchanged stable conduction abnormalities e.g., right bundle branch block, or any other finding which does not significantly impact mortality.
10. Pre-existing co-morbid condition(s) preventing outcome assessments, e.g. disease or condition that would prevent ability to transfer and walk for 6 minutes, prior to confirmed COVID-19 diagnosis (assisted walking devices are acceptable)
11. As a result of the medical review and screening investigation, the Principal Investigator considers the patient unfit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ampio Pharmaceuticals, Englewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Ampion
  Ampion: Inhaled nebulized Ampion (8 mL) administered four times daily, every four to six hours, for five days.
- Control: Placebo
  Placebo: Inhaled nebulized saline (8 mL) administered four times daily, every four to six hours, for five days.
Period: Overall Study
Arm/Group | Active | Control
Started | 16 | 16
Completed | 14 | 13
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Compliance | 1 | 1
Not completed — Incorrectly Randomized followed for Safety | 0 | 1
Not completed — Screen Failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (11.9) | 55.1 (13.7) | 52.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.6 (7.4) | 34.1 (7.0) | 33.4 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment Emergent Adverse Events of Ampion Compared to Placebo
Description: Number of subjects with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of treatment of inhalation Ampion compared to Placebo. AEs were assessed based on symptoms as a severity rating of mild, moderate, or severe. The relationship between AE and study drug was determined as either unrelated, possibly related, or related. SAEs are defined as resulting death, life threatening, requires prolonged hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect.
Time Frame: Baseline to Day 28
Population: Safety Population - one participant from the Active population was randomized, but did not receive treatment and thus was not included from the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 15 | 16
Participants
  Subjects with Treatment Emergent Adverse Events (TEAE's) | 5 | 9
  Subjects with Study Drug Related TEAE's | 3 | 5
  Subjects with Moderate or Severe TEAE's | 1 | 5
  Subjects with SAE's | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Day 60
Description: Patients were followed for the occurrence of Adverse Events for 60 days following the first dose of study medication. One participant from the Active population was randomized, but did not receive treatment and thus was not included from the safety population.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 8/15 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=15) | Control (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT04880161/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04880161/SAP_001.pdf